CLINICAL TRIAL: NCT02948582
Title: Randomized, Placebo-Controlled, Double-Blind, Dose Ranging, Single-Dose, 6-Way Crossover Study to Assess Safety, Efficacy and Pharmacokinetics of EP-101 Using eFlow Nebuliser in Patients With COPD
Brief Title: Assessment of the Safety and Ability of a Once-a-day Dose of an Orally Inhaled Medicine [i.e., Glycopyrrolate Inhalation Solution = GIS] to Improve Airflow in the Lungs When Delivered Using an eFlow Nebulizer in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunovion Respiratory Development Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: EP-101-02; 2010-018987-17 (EudraCT Number)
Record Dates: First submitted 2016-10-26; First posted 2016-10-28 (Estimated); Results first posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Emphysema; Chronic bronchitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Glycopyrrolate Inhalation Solution12.5μg (Experimental): Glycopyrrolate Inhalation Solution12.5μg via e-flow nebulizer, once daily
  Interventions: Drug: Glycopyrrolate Inhalation Solution12.5μg
- Glycopyrrolate Inhalation Solution 50μg (Experimental): Glycopyrrolate Inhalation Solution 50mg via e-flow nebulizer, once daily
  Interventions: Drug: Glycopyrrolate Inhalation Solution 50μg
- Glycopyrrolate Inhalation Solution 100μg (Experimental): Glycopyrrolate Inhalation Solution 100μg via e-flow nebulizer, once daily
  Interventions: Drug: Glycopyrrolate Inhalation Solution 100μg
- Glycopyrrolate Inhalation Solution 200μg (Experimental): Glycopyrrolate Inhalation Solution 200μg via e-flow nebulizer, once daily
  Interventions: Drug: Glycopyrrolate Inhalation Solution 200μg
- Glycopyrrolate Inhalation Solution 400μg (Experimental): Glycopyrrolate Inhalation Solution 400μg via e-flow nebulizer, once daily
  Interventions: Drug: Glycopyrrolate Inhalation Solution 400μg
- Placebo 0.5mL (Placebo Comparator): Placebo 0.5mL via e-flow nebulizer, once daily
  Interventions: Drug: Placebo 0.5mL

INTERVENTIONS:
Drug: Glycopyrrolate Inhalation Solution12.5μg — Glycopyrrolate Inhalation Solution12.5μg via eFlow, once daily
  Other Names: GIS
  Arms: Glycopyrrolate Inhalation Solution12.5μg
Drug: Glycopyrrolate Inhalation Solution 50μg — Glycopyrrolate Inhalation Solution 50μg via eFlow, once daily
  Other Names: GIS
  Arms: Glycopyrrolate Inhalation Solution 50μg
Drug: Glycopyrrolate Inhalation Solution 100μg — Glycopyrrolate Inhalation Solution 100μg via eFlow, once daily
  Other Names: GIS
  Arms: Glycopyrrolate Inhalation Solution 100μg
Drug: Glycopyrrolate Inhalation Solution 200μg — Glycopyrrolate Inhalation Solution 200μg via eFlow, once daily
  Other Names: GIS
  Arms: Glycopyrrolate Inhalation Solution 200μg
Drug: Glycopyrrolate Inhalation Solution 400μg — Glycopyrrolate Inhalation Solution 400μg via eFlow, once daily
  Other Names: GIS
  Arms: Glycopyrrolate Inhalation Solution 400μg
Drug: Placebo 0.5mL — Placebo 0.5mL via eFlow, once daily
  Other Names: Placebo
  Arms: Placebo 0.5mL

SUMMARY:
The study assessed the safety and ability of an orally inhaled medicine [i.e., Glycopyrrolate Inhalation Solution = GIS] to improve airflow in the lungs when delivered using an eFlow nebulizer in 42 patients with Chronic Obstructive Pulmonary Disease (COPD). Each patient randomly received several, single doses of GIS, or placebo, separated by approximately 1 to 2 weeks. After the dose was given, lung airflow was measured over 24 hours and blood was collected to measure how much GIS was in the bloodstream. The study was conducted to find the once-a- day GIS dose that produced the highest improvement in lung airflow using the eFlow nebulizer.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 40 through 75 years, inclusive
2. A clinical diagnosis of COPD according to the GOLD guidelines
3. Current smokers or ex-smokers with at least 10 pack-year smoking history (e.g., at least 1 pack/day for 10
4. Post-bronchodilator FEV1 30-70% of predicted normal at the Screening Visit
5. Post-bronchodilator FEV1/FVC ratio < 0.70 at the Screening Visit
6. Improvement in FEV1 >12% and 150 mL following inhalation of ipratropium bromide at the Screening Visit
7. Ability to perform reproducible spirometry according to the ATS/ERS guidelines
8. Willing to stay at the study site for approximately 30 hours on each treatment visit
9. Willing and able to provide written informed consent

Exclusion Criteria:

1. Females who are pregnant or lactating at the Screening Visit, or if of childbearing potential not using one of the following acceptable means of birth control throughout the study:

   * Abstinence
   * Post-menopausal for at least two years
   * Surgically sterile (i.e., tubal ligation, hysterectomy)
   * Oral contraceptives (taken for at least one month prior to the Screening Visit)
   * Approved implantable or injectable contraceptives (e.g., Norplant®, Depo-Provera® or equivalent)
   * Barrier methods (e.g., condoms with spermicide)
   * Intrauterine device (i.e., IUD)
   * Vasectomy of male partner
   * Non-heterosexual life style
2. Current evidence or recent history of any clinically significant disease (other than COPD) or abnormality in the opinion of the Investigator that would put the subject at risk or which would compromise the quality of the study data; including but not limited to cardiovascular disease, myocardial infarction, cardiac failure, uncontrolled hypertension, life-threatening arrhythmias, uncontrolled diabetes, neurologic or neuromuscular disease, liver disease, gastrointestinal disease or electrolyte abnormalities
3. Recent history of hospitalization due to an exacerbation of airway disease within 3 months or need for increased treatments for COPD within 6 weeks prior to the Screening Visit
4. Primary diagnosis of asthma
5. Prior lung volume reduction surgery or history of chest/lung irradiation
6. Regular use of daily oxygen therapy
7. Use of systemic (eg, intramuscular or intravenous) steroids within 3 months prior to the Screening Visit
8. Respiratory tract infection within 6 weeks prior to the Screening Visit
9. History of tuberculosis, bronchiectasis or other non- specific pulmonary disease
10. History of urinary retention or bladder neck obstruction type symptoms
11. History of narrow-angle glaucoma
12. Clinically significant abnormal ECG
13. Positive Hepatitis B surface antigen or positive Hepatitis C antibody
14. Positive screening test for HIV antibodies
15. Current or recent history (previous 12 months) of excessive use or abuse of alcohol
16. Current evidence or history of abusing legal drugs or use of illegal drugs or substances
17. Donation of 450 mL of blood within 8 weeks of the Screening Visit
18. History of hypersensitivity or intolerance to aerosol medications
19. Participation in another investigational drug study was received within 30 days prior to the Screening Visit

Ages: 40 Years to 75 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Tutuncu, MD, PhD, Study Chair — Elevation Pharmaceuticals, Inc., (now known as Sunovion Respriatory Developement Inc.)

REFERENCES:
- [Result] Leaker BR, Barnes PJ, Jones CR, Tutuncu A, Singh D. Efficacy and safety of nebulized glycopyrrolate for administration using a high efficiency nebulizer in patients with chronic obstructive pulmonary disease. Br J Clin Pharmacol. 2015 Mar;79(3):492-500. doi: 10.1111/bcp.12517. PMID 25243340

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled subjects were randomized. all randomized subjects received at least one dose of study medication
Groups:
- Treatment Group 1: subjects received placebo, glycopyrrolate 400mcg, glycopyrrolate 50 mcg, glycopyrrolate 12.5 mcg, glycoyrrolate 200mcg, or glycopryrrolate 100mcg
- Treatment Group 2: subjects received glycopyrrolate 12.5 mcg, glycopyrrolate 50 mcg, glycopryrrolate 100mcg, placebo, glycopyrrolate 200mcg, glycoyrrolate 400mcg, or placebo
- Treatment Group 3: subjects received glycopyrrolate 50 mcg, Placebo, glycopyrrolate 200 mcg, glycopryrrolate 100mcg, glycopyrrolate 12.5mcg, or glycoyrrolate 400mcg
- Treatment Group 4: subjects received glycopyrrolate 100 mcg, glycopyrrolate 200 mcg, glycopryrrolate 400mcg, placebo, glycopyrrolate 50mcg, or glycoyrrolate 12.5mcg
- Treatment Group 5: subjects received glycopyrrolate 200 mcg, glycopyrrolate 12.5 mcg, placebo, glycopryrrolate 400mcg, placebo, glycopyrrolate 100mcg, or glycoyrrolate 50mcg
- Treatment Group 6: subjects received glycopyrrolate 400 mcg, glycopyrrolate 100 mcg, glycopryrrolate 12.5mcg, glycopyrrolate 50mcg, placebo or glycoyrrolate 200mcg
Period: Treatment Period 1
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Started | 7 | 7 | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Started | 7 | 7 | 7 | 7 | 7 | 7
Completed | 7 | 5 | 7 | 7 | 7 | 6
Not Completed | 0 | 2 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1
Period: Treatment Period 2
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Started | 7 | 5 | 7 | 7 | 7 | 6
Completed | 7 | 5 | 7 | 7 | 7 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Started | 7 | 5 | 7 | 7 | 7 | 6
Completed | 7 | 4 | 7 | 6 | 7 | 6
Not Completed | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Not completed — personal reasons | 0 | 0 | 0 | 1 | 0 | 0
Period: Treatment Period 3
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Started | 7 | 4 | 7 | 6 | 7 | 6
Completed | 7 | 4 | 7 | 6 | 7 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 3
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Started | 7 | 4 | 7 | 6 | 7 | 6
Completed | 7 | 4 | 7 | 6 | 7 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 4
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Started | 7 | 4 | 7 | 6 | 7 | 6
Completed | 7 | 4 | 7 | 6 | 7 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 4
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Started | 7 | 4 | 7 | 6 | 7 | 6
Completed | 6 | 4 | 6 | 6 | 7 | 6
Not Completed | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 0 | 0
Period: Treatment Period 5
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Started | 6 | 4 | 6 | 6 | 7 | 6
Completed | 6 | 4 | 6 | 6 | 7 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 5
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Started | 6 | 4 | 6 | 6 | 7 | 6
Completed | 6 | 4 | 6 | 6 | 7 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 6
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Started | 6 | 4 | 6 | 6 | 7 | 6
Completed | 6 | 4 | 6 | 6 | 7 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Wshout Period 6
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Started | 6 | 4 | 6 | 6 | 7 | 6
Completed | 6 | 4 | 6 | 6 | 7 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat population same as safety population -not full analysis set
Groups:
- Total Participants: Intent to treat population same as safety population -not full analysis set
Arm/Group | Total Participants
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (6.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 41
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 42

OUTCOME MEASURES:

1. Primary Outcome: Trough FEV1 (Change From Baseline)
Description: Spirometry measurements were conducted in accordance with the current ATS/ERS 2005 guidelines.
  Trough FEV1 was defined as the mean of FEV1 values obtained at 23 hours 30 minutes and 24 hours post-dose of each Treatment Visit.
Time Frame: 24hr post dose
Population: All subjects who received at least one dose of study medication and had at least one postbaseline efficacy measurement (FEV1) were included in the intent-to-treat analysis.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Glycopyrrolate Inhalation Solution12.5μg | Glycopyrrolate Inhalation Solution 50μg | Glycopyrrolate Inhalation Solution 100μg | Glycopyrrolate Inhalation Solution 200μg | Glycopyrrolate Inhalation Solution 400μg | Placebo 0.5mL
Number analyzed (Participants) | 38 | 38 | 37 | 37 | 37 | 37
liters | -0.093 (0.1189) | 0.0114 (0.1308) | 0.0447 (0.1548) | 0.0542 (0.1779) | 0.0292 (0.1468) | -0.0612 (0.1233)
Statistical Analysis 1: Comparison: Glycopyrrolate Inhalation Solution12.5μg vs Placebo 0.5mL; An analysis of covariance was used with change from baseline in trough FEV1 as the response, with factors for center, treatment, period, sequence, baseline FEV1 as a covariate and a random effect for subject nested within sequence. A sample size of 34 subjects (42 with dropouts) provides 80% power to detect a 0.14L difference in mean change trough FEV1 between 2 groups at an alpha of 0.05 using a 2-tailed t-test and assuming a common standard deviation for change in trough FEV1 of 0.2; Test type: Superiority; p = 0.1257, least squares mean; least squares mean = 0.033, 95% CI 2-sided [-0.009 to 0.075]
Statistical Analysis 2: Comparison: Glycopyrrolate Inhalation Solution 50μg vs Placebo 0.5mL; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0008, least squares mean; least squares mean = 0.072, 95% CI 2-sided [0.030 to 0.113]
Statistical Analysis 3: Comparison: Glycopyrrolate Inhalation Solution 100μg vs Placebo 0.5mL; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, least squares mean; least squares mean = 0.102, 95% CI 2-sided [0.061 to 0.144]
Statistical Analysis 4: Comparison: Glycopyrrolate Inhalation Solution 200μg vs Placebo 0.5mL; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, least squares mean; least squares mean = 0.108, 95% CI 2-sided [0.066 to 0.150]
Statistical Analysis 5: Comparison: Glycopyrrolate Inhalation Solution 400μg vs Placebo 0.5mL; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, least squares mean; least squares mean = 0.098, 95% CI 2-sided [0.056 to 0.140]

2. Primary Outcome: Standardized FEV1AUC0-12 Area Under the FEV1 Curve From 0 to 12 Hours Post-dose ( Actual and Change From Baseline).
Description: Spirometry measurements were conducted in accordance with the current ATS/ERS 2005 guidelines.. The standardized actual FEV1 AUC(0-12) was calculated using the trapezoidal rule divided by the actual hours from the first FEV1 to the last FEV1 in the interval. Standardized change from baseline FEV1 AUC(0-12) was also calculated similarly, using the change from pre-dose FEV1.
Time Frame: 0-12h post dose
Population: All subjects who received at least one dose of study medication and had at least one postbaseline efficacy measurement (FEV1) were included in the intent to treat analysis
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Glycopyrrolate Inhalation Solution12.5μg | Glycopyrrolate Inhalation Solution 50μg | Glycopyrrolate Inhalation Solution 100μg | Glycopyrrolate Inhalation Solution 200μg | Glycopyrrolate Inhalation Solution 400μg | Placebo 0.5mL
Number analyzed (Participants) | 39 | 38 | 37 | 37 | 37 | 37
liters
  actual standardized FEV1 AUC0_12 | 1.259 (0.409) | 1.311 (0.422) | 1.335 (0.394) | 1.374 (0.391) | 1.390 (0.423) | 1.180 (0.427)
  change from baseline standardized FEV1 AUC0_12 | 0.055 (0.113) | 0.126 (0.112) | 0.136 (0.134) | 0.184 (0.134) | 0.170 (0.110) | -0.024 (0.095)
Statistical Analysis 1: Comparison: Glycopyrrolate Inhalation Solution12.5μg vs Placebo 0.5mL; An analysis of covariance was used with change from baseline in standardized FEV1 AUC0_12 as the response, with factors for center, treatment, period, sequence, baseline FEV1 as a covariate and a random effect for subject nested within sequence; Test type: Superiority; p < 0.0001, least squares mean; least squares mean = 0.086, 95% CI 2-sided [0.050 to 0.123]
Statistical Analysis 2: Comparison: Glycopyrrolate Inhalation Solution 50μg vs Placebo 0.5mL; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, least squares mean; least squares mean = 0.151, 95% CI 2-sided [0.114 to 0.187]
Statistical Analysis 3: Comparison: Glycopyrrolate Inhalation Solution 100μg vs Placebo 0.5mL; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, least squares mean; least squares mean = 0.156, 95% CI 2-sided [0.120 to 0.193]
Statistical Analysis 4: Comparison: Glycopyrrolate Inhalation Solution 200μg vs Placebo 0.5mL; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, least squares mean; least squares mean = 0.202, 95% CI 2-sided [0.165 to 0.239]
Statistical Analysis 5: Comparison: Glycopyrrolate Inhalation Solution 400μg vs Placebo 0.5mL; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, least squares mean; least squares mean = 0.199, 95% CI 2-sided [0.162 to 0.235]

3. Primary Outcome: Standardized FEV1AUC12-24 Area Under the FEV1 Curve From 12 to 24 Hours Post- Dose (Actual and Change From Baseline).
Description: Spirometry measurements were conducted in accordance with the current ATS/ERS 2005 guidelines. The standardized actual FEV1 AUC(12-24) was calculated using the trapezoidal rule divided by the actual hours from the first FEV1 to the last FEV1 in the interval. Standardized change from baseline FEV1 AUC(12-24) was also calculated similarly, using the change from pre-dose FEV1.
Time Frame: 12-24h post dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Glycopyrrolate Inhalation Solution12.5μg | Glycopyrrolate Inhalation Solution 50μg | Glycopyrrolate Inhalation Solution 100μg | Glycopyrrolate Inhalation Solution 200μg | Glycopyrrolate Inhalation Solution 400μg | Placebo 0.5mL
Number analyzed (Participants) | 39 | 38 | 37 | 37 | 37 | 37
liters
  acutal standardized FEV1 AUC0_12 | 1.165 (0.377) | 1.203 (0.404) | 1.227 (0.369) | 1.253 (0.346) | 1.259 (0.396) | 1.123 (0.392)
  change from baseline standardized FEV1 AUC0_12 | -0.038 (0.132) | 0.018 (0.135) | 0.028 (0.138) | 0.063 (0.178) | 0.039 (0.135) | -0.082 (0.120)
Statistical Analysis 1: Comparison: Glycopyrrolate Inhalation Solution12.5μg vs Placebo 0.5mL; An analysis of covariance was used with change from baseline in standardized FEV1 AUC12_24 as the response, with factors for center, treatment, period, sequence, baseline FEV1 as a covariate and a random effect for subject nested within sequence; Test type: Superiority; p = 0.0028, least squares mean; least squares mean = 0.058, 95% CI 2-sided [0.021 to 0.095]
Statistical Analysis 2: Comparison: Placebo 0.5mL; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, least squares mena; least squares mean = 0.100, 95% CI 2-sided [0.063 to 0.137]
Statistical Analysis 3: Comparison: Glycopyrrolate Inhalation Solution 100μg vs Placebo 0.5mL; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, least squares mean; least squares mean = 0.105, 95% CI 2-sided [0.068 to 0.142]
Statistical Analysis 4: Comparison: Glycopyrrolate Inhalation Solution 200μg vs Placebo 0.5mL; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, least squares mean; least squares mean = 0.135, 95% CI 2-sided [0.098 to 0.173]
Statistical Analysis 5: Comparison: Placebo 0.5mL; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, least squares mean; least squares mean = 0.128, 95% CI 2-sided [0.091 to 0.166]

4. Primary Outcome: Standardized FEV1 AUC0-24 Area Under the FEV1 Curve From 0 to 24 Hours Post-dose (Actual and Change Baseline)
Description: Spirometry measurements were conducted in accordance with the current ATS/ERS 2005 guidelines. . The standardized actual FEV1 AUC(0-24) was calculated using the trapezoidal rule divided by the actual hours from the first FEV1 to the last FEV1 in the interval. Standardized change from baseline FEV1 AUC(0-24) was also calculated similarly, using the change from pre-dose FEV1.
Time Frame: 0 to 24h
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Glycopyrrolate Inhalation Solution12.5μg | Glycopyrrolate Inhalation Solution 50μg | Glycopyrrolate Inhalation Solution 100μg | Glycopyrrolate Inhalation Solution 200μg | Glycopyrrolate Inhalation Solution 400μg | Placebo 0.5mL
Number analyzed (Participants) | 39 | 38 | 37 | 37 | 37 | 37
liters
  Actual standardized FEV1 AUC0_12 | 1.212 (0.391) | 1.257 (0.411) | 1.281 (0.379) | 1.313 (0.364) | 1.325 (0.407) | 1.151 (0.408)
  change from baseline standardized FEV1 AUC0_12 | 0.009 (0.114) | 0.072 (0.115) | 0.082 (0.128) | 0.123 (0.146) | 0.105 (0.113) | -0.053 (0.102)

5. Primary Outcome: Peak FEV1 (Change From Baseline and Percent Change)
Description: spirometry measurements were conducted in accordance with the current ATS/ERS 2005 guidelines. . The peak FEV1 was defined as the highest post-dose FEV1 value within 4 hrs after the dose. Percent change from baseline was calculated as 100 times the difference of peak FEV1 minus baseline FEV1 divided by baseline FEV1.
Time Frame: 0-4h post dose
Population: all subjects who received at least one dose of study medication and have at least one post baseline efficacy measurement were included in the efficacy population
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Glycopyrrolate Inhalation Solution12.5μg | Glycopyrrolate Inhalation Solution 50μg | Glycopyrrolate Inhalation Solution 100μg | Glycopyrrolate Inhalation Solution 200μg | Glycopyrrolate Inhalation Solution 400μg | Placebo 0.5mL
Number analyzed (Participants) | 39 | 38 | 37 | 37 | 37 | 37
liters
  Change from baseline | 0.165 (0.113) | 0.229 (0.113) | 0.260 (0.151) | 0.292 (0.120) | 0.272 (0.125) | 0.061 (0.102)
  percent change from baseline | 15.30 (11.37) | 21.05 (11.87) | 24.14 (20.69) | 26.73 (12.56) | 25.44 (15.10) | 5.24 (8275)

6. Secondary Outcome: Cmax; Maximum Observed Plasma Concentration
Description: Pk parameters are calculated from glycopyrrolate plasma concentration analysed from serial blood samples collected between 0 and 12 hr
Time Frame: 0 to 12 hour
Population: All subjects who received at least one dose of EP-101 and who have sufficient blood samples taken to obtain a plasma concentration by time profile and have no major protocol violations were included in the PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Glycopyrrolate Inhalation Solution12.5μg | Glycopyrrolate Inhalation Solution 50μg | Glycopyrrolate Inhalation Solution 100μg | Glycopyrrolate Inhalation Solution 200μg | Glycopyrrolate Inhalation Solution 400μg
Number analyzed (Participants) | 2 | 13 | 12 | 12 | 13
pg/mL | 59.25 (78.49) | 74.48 (62.24) | 144.58 (52.53) | 316.05 (48.35) | 504.93 (55.67)

7. Secondary Outcome: Tmax; Time to Maximum Observed Plasma Concentration
Description: as for outcome 6
Time Frame: 0 to 12 hours
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | Glycopyrrolate Inhalation Solution12.5μg | Glycopyrrolate Inhalation Solution 50μg | Glycopyrrolate Inhalation Solution 100μg | Glycopyrrolate Inhalation Solution 200μg | Glycopyrrolate Inhalation Solution 400μg
Number analyzed (Participants) | 2 | 13 | 12 | 12 | 12
hours | 0.165 [0.150 to 0.180] | 0.320 [.0150 to 0.350] | 0.260 [0.150 to 0.330] | 0.275 [0.150 to 0.380] | 0.180 [0.150 to 0.320]

8. Secondary Outcome: t1/2; Plasma Half-life
Description: as for outcome 6
Time Frame: 0 to 12 hour
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Glycopyrrolate Inhalation Solution12.5μg | Glycopyrrolate Inhalation Solution 50μg | Glycopyrrolate Inhalation Solution 100μg | Glycopyrrolate Inhalation Solution 200μg | Glycopyrrolate Inhalation Solution 400μg
Number analyzed (Participants) | 0 | 2 | 4 | 7 | 6
hours |  | 0.8949 (2.3707) | 3.0137 (50.7557) | 3.1663 (45.4839) | 4.1238 (63.5353)

9. Secondary Outcome: AUC0-t; Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Measurable Drug Concentration.
Description: as for outcome 6
Time Frame: 0 to 12 hour
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg.h/ml
Arm/Group | Glycopyrrolate Inhalation Solution12.5μg | Glycopyrrolate Inhalation Solution 50μg | Glycopyrrolate Inhalation Solution 100μg | Glycopyrrolate Inhalation Solution 200μg | Glycopyrrolate Inhalation Solution 400μg
Number analyzed (Participants) | 2 | 13 | 12 | 12 | 13
pg.h/ml | 135.87 (209.27) | 67.18 (143.22) | 237.80 (98.45) | 677.24 (66.34) | 1481.36 (82.17)

10. Secondary Outcome: AUC0-inf Area Under the Plasma Concentration-time Curve From Time Zero to Infinity
Description: as for outcome 6
Time Frame: 0 to 12 hour
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg.h/ml
Arm/Group | Glycopyrrolate Inhalation Solution12.5μg | Glycopyrrolate Inhalation Solution 50μg | Glycopyrrolate Inhalation Solution 100μg | Glycopyrrolate Inhalation Solution 200μg | Glycopyrrolate Inhalation Solution 400μg
Number analyzed (Participants) | 0 | 2 | 4 | 7 | 6
pg.h/ml |  | 246.84 (37.49) | 634.65 (34.28) | 772.59 (26.30) | 1367.76 (76.70)

11. Secondary Outcome: Number of Subjects Who Died, Number of Subjects With Treatment Emergent SAEs, Number of Subjects Who Discontinued Due to AE
Description: AE's are defined as existing conditions which worsen or events which occur during the course of the clinical trial after treatment
Time Frame: Day 69 (includes dosing Day 1, washout Day 12, safety follow up Day 69)
Population: all subjects who received at least one dose of study drug were included in the safety analysis
Measure: Number; unit: participants
Arm/Group | Glycopyrrolate Inhalation Solution12.5μg | Glycopyrrolate Inhalation Solution 50μg | Glycopyrrolate Inhalation Solution 100μg | Glycopyrrolate Inhalation Solution 200μg | Glycopyrrolate Inhalation Solution 400μg | Placebo 0.5mL
Number analyzed (Participants) | 39 | 38 | 37 | 37 | 37 | 37
participants
  subjects who died | 0 | 0 | 0 | 0 | 0 | 0
  subjects with treatment emergent SAEs | 0 | 0 | 1 | 0 | 0 | 0
  Subjects whodiscontinued due to an AE | 2 | 2 | 2 | 0 | 0 | 0
  subjects with treatment emergent AEs | 16 | 14 | 17 | 15 | 13 | 14

12. Secondary Outcome: Number of Subjects With Clinically Significant Abnormal Vital Signs Reported During the Study
Description: Vital signs were measured at screening and at each Treatment Visit pre-dose (within 30 minutes prior to dose); post-dose at 30 minutes and 1, 2, 4, 8, 12 and 24 hours; and then at the post study assessment.
Time Frame: 0-24 h
Population: all subjects who received at least one does of study drug were included in the safety analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Glycopyrrolate Inhalation Solution12.5μg | Glycopyrrolate Inhalation Solution 50μg | Glycopyrrolate Inhalation Solution 100μg | Glycopyrrolate Inhalation Solution 200μg | Glycopyrrolate Inhalation Solution 400μg | Placebo 0.5mL
Number analyzed (Participants) | 39 | 38 | 37 | 37 | 37 | 37
Participants | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Clinically Significant Abnormal Laboratory Results Reported During the Study
Description: Clinical safety lab parameters were collected at screening and at the post study assessment. Any laboratory values that were out of range of normal reference values were evaluated by the Investigators.
Time Frame: Day -14, Day 69
Population: all subjects who received at least one dose of study drug were included in the safety analysis
Measure: Number; unit: number of events
Arm/Group | Glycopyrrolate Inhalation Solution12.5μg | Glycopyrrolate Inhalation Solution 50μg | Glycopyrrolate Inhalation Solution 100μg | Glycopyrrolate Inhalation Solution 200μg | Glycopyrrolate Inhalation Solution 400μg | Placebo 0.5mL
Number analyzed (Participants) | 39 | 38 | 37 | 37 | 37 | 37
number of events | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Subjects With Clinically Significant ECG Parameters Reported During the Study
Description: ECGs were recorded at screening and at each study treatment visit pre-dose (within 30 minutes prior to dose); post-dose at 30 minutes and 1, 2, 4, 8, 12 and 24 hours; and then at the post study assessment.
Time Frame: 0 to 24h
Population: all subjects who received at least one dose of study drug were included in the safety analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Glycopyrrolate Inhalation Solution12.5μg | Glycopyrrolate Inhalation Solution 50μg | Glycopyrrolate Inhalation Solution 100μg | Glycopyrrolate Inhalation Solution 200μg | Glycopyrrolate Inhalation Solution 400μg | Placebo 0.5mL
Number analyzed (Participants) | 39 | 38 | 37 | 37 | 37 | 37
Participants | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Percentage of Subjects With Treatment Emergent AEs
Description: as for outcome 11
Time Frame: Day 69 (includes dosing Day 1, washout Day 12, safety follow up Day 69)
Population: all subjects who received at least one dose of study drug were included in the safety analysis
Measure: Number; unit: percentage of participants
Arm/Group | Glycopyrrolate Inhalation Solution12.5μg | Glycopyrrolate Inhalation Solution 50μg | Glycopyrrolate Inhalation Solution 100μg | Glycopyrrolate Inhalation Solution 200μg | Glycopyrrolate Inhalation Solution 400μg | Placebo 0.5mL
Number analyzed (Participants) | 39 | 38 | 37 | 37 | 37 | 37
percentage of participants | 41.0 | 36.8 | 45.9 | 40.5 | 35.1 | 37.8

ADVERSE EVENTS:
Time Frame: 0-69 days
Description: AEs are defined as existing conditions which worsen or events which occur during the course of the clinical trial after treatment
Arm/Group | Glycopyrrolate Inhalation Solution12.5μg | Glycopyrrolate Inhalation Solution 50μg | Glycopyrrolate Inhalation Solution 100μg | Glycopyrrolate Inhalation Solution 200μg | Glycopyrrolate Inhalation Solution 400μg | Placebo 0.5mL
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/38 | 1/37 | 0/37 | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 13/39 | 9/38 | 10/37 | 10/37 | 10/37 | 10/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glycopyrrolate Inhalation Solution12.5μg (N=39) | Glycopyrrolate Inhalation Solution 50μg (N=38) | Glycopyrrolate Inhalation Solution 100μg (N=37) | Glycopyrrolate Inhalation Solution 200μg (N=37) | Glycopyrrolate Inhalation Solution 400μg (N=37) | Placebo 0.5mL (N=37)
groin pain (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glycopyrrolate Inhalation Solution12.5μg (N=39) | Glycopyrrolate Inhalation Solution 50μg (N=38) | Glycopyrrolate Inhalation Solution 100μg (N=37) | Glycopyrrolate Inhalation Solution 200μg (N=37) | Glycopyrrolate Inhalation Solution 400μg (N=37) | Placebo 0.5mL (N=37)
skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
headache (Nervous system disorders) | 6 (7) | 5 (6) | 5 (8) | 7 (9) | 6 (8) | 4 (5)
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 5 (5) | 3 (3) | 3 (4) | 5 (5)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (2) | 1 (1) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.